CLINICAL TRIAL: NCT02959450
Title: Design and Implementation of a Nutritional Intervention in Patients With Oropharyngeal Dysphagia. Compared With Traditional Practice: Randomized Clinical Trial, Simple Blind
Brief Title: Design and Implementation of a Nutritional Intervention in Patients With Oropharyngeal Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Aurora Elizabeth Serralde Zúñiga, MD, PhD, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1557
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Oropharyngeal Dysphagia
Keywords: Nutritional Intervention in Oropharyngeal Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified consistency and volume diet (Experimental): Modified consistency diet, with a certain viscosity and controlled volume. The nectar consistency had a viscosity of 51 to 350 centiPoises (cP) and the pudding consistency menus with a higher viscosity at 1,750 cP.
  Interventions: Dietary Supplement: Modified consistency and volume diet
- Control Group (No Intervention): Standard treatment consisting of a modified consistency diet with adequate intake of energy and protein and general recommendations on diet prescribed by the treating physician

INTERVENTIONS:
Dietary Supplement: Modified consistency and volume diet — Modified consistency diet, with a certain viscosity and controlled volume, which was designed from recommendations based on the review of different studies. A Chef and a Nutritionist developed and determined the viscosity of the menus with a Brookfield Viscometer (model RV). All the menus were prepared and evaluated at the Food Technology Department of this Institute to achieve the viscosity required with a food thickener. The nectar consistency had a viscosity of 51 to 350 centiPoises (cP) and the pudding consistency menus with a higher viscosity at 1,750 cP. The patient and/or their caregivers in the intervention group must attend to a training workshop to explain how to use the food thickener.
  Arms: Modified consistency and volume diet

SUMMARY:
The purpose of this trial is to design, implement and evaluate the effect of a nutritional intervention in patients with Oropharyngeal Dysphagia on body composition and oral intake of energy and protein.

DETAILED DESCRIPTION:
Oropharyngeal Dysphagia causes complications that compromise the efficacy and security of deglutition. An inefficacy deglutition increases the risk of malnutrition and/or dehydration. On the other hand, unsafe deglutition requires more time to complete the oral preparation of the bolus, which can leave residues in the mouth that can then lead to penetration of small food particles into the respiratory tract. These tracheobronchial aspirations cause aspiration pneumonia in 50% of cases, with 50% of mortality rate.

Despite the enormous impact of Oropharyngeal Dysphagia in functional capacity and quality of life, this problem is underestimated and underdiagnosed as a major cause of nutritional and pulmonary complications that generate more material and human resources. There are few studies evaluating the effect of a nutritional intervention on recovery in swallowing ability or improvement of nutritional status.

The purpose of this trial is to design a nutritional intervention with modified texture foods to increase viscosity (measured accurately) according to the patient's requirements, also assess if the intervention has a positive effect on the swallowing ability, calorie and protein oral intake and nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Oropharyngeal Dysphagia.
* Patients who have primary caregiver.
* Agreeing to participate in the study.

Exclusion Criteria:

* Critically ill patients.
* Chronic kidney disease with Glomerular Filtration Rate <30 ml / min or in renal replacement therapy
* Liver failure.
* Cancer with active radiotherapy or chemotherapy treatment.
* Patients who are participating in another study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2015-05; Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aurora E Serralde-Zúñiga, MD, PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Clave P, Verdaguer A, Arreola V. [Oral-pharyngeal dysphagia in the elderly]. Med Clin (Barc). 2005 May 21;124(19):742-8. doi: 10.1157/13075447. No abstract available. Spanish. PMID 15919036
- [Result] Roden DF, Altman KW. Causes of dysphagia among different age groups: a systematic review of the literature. Otolaryngol Clin North Am. 2013 Dec;46(6):965-87. doi: 10.1016/j.otc.2013.08.008. Epub 2013 Oct 12. PMID 24262954
- [Result] Clave P, Terre R, de Kraa M, Serra M. Approaching oropharyngeal dysphagia. Rev Esp Enferm Dig. 2004 Feb;96(2):119-31. doi: 10.4321/s1130-01082004000200005. No abstract available. English, Spanish. PMID 15255021
- [Result] Clave P, Arreola V, Romea M, Medina L, Palomera E, Serra-Prat M. Accuracy of the volume-viscosity swallow test for clinical screening of oropharyngeal dysphagia and aspiration. Clin Nutr. 2008 Dec;27(6):806-15. doi: 10.1016/j.clnu.2008.06.011. Epub 2008 Sep 11. PMID 18789561
- [Result] Wallace KL, Middleton S, Cook IJ. Development and validation of a self-report symptom inventory to assess the severity of oral-pharyngeal dysphagia. Gastroenterology. 2000 Apr;118(4):678-87. doi: 10.1016/s0016-5085(00)70137-5. PMID 10734019
- [Result] Belafsky PC, Mouadeb DA, Rees CJ, Pryor JC, Postma GN, Allen J, Leonard RJ. Validity and reliability of the Eating Assessment Tool (EAT-10). Ann Otol Rhinol Laryngol. 2008 Dec;117(12):919-24. doi: 10.1177/000348940811701210. PMID 19140539
- [Result] Burgos R, Sarto B, Segurola H, Romagosa A, Puiggros C, Vazquez C, Cardenas G, Barcons N, Araujo K, Perez-Portabella C. [Translation and validation of the Spanish version of the EAT-10 (Eating Assessment Tool-10) for the screening of dysphagia]. Nutr Hosp. 2012 Nov-Dec;27(6):2048-54. doi: 10.3305/nh.2012.27.6.6100. Spanish. PMID 23588456
- [Result] Aviv JE, Sataloff RT, Cohen M, Spitzer J, Ma G, Bhayani R, Close LG. Cost-effectiveness of two types of dysphagia care in head and neck cancer: a preliminary report. Ear Nose Throat J. 2001 Aug;80(8):553-6, 558. PMID 11523474
- [Result] Carrion S, Cabre M, Monteis R, Roca M, Palomera E, Serra-Prat M, Rofes L, Clave P. Oropharyngeal dysphagia is a prevalent risk factor for malnutrition in a cohort of older patients admitted with an acute disease to a general hospital. Clin Nutr. 2015 Jun;34(3):436-42. doi: 10.1016/j.clnu.2014.04.014. Epub 2014 May 9. PMID 24882372
- [Result] Finestone HM, Greene-Finestone LS. Rehabilitation medicine: 2. Diagnosis of dysphagia and its nutritional management for stroke patients. CMAJ. 2003 Nov 11;169(10):1041-4. PMID 14609974
- [Result] Jonsson AC, Lindgren I, Norrving B, Lindgren A. Weight loss after stroke: a population-based study from the Lund Stroke Register. Stroke. 2008 Mar;39(3):918-23. doi: 10.1161/STROKEAHA.107.497602. Epub 2008 Jan 31. PMID 18239168
- [Result] Brynningsen PK, Damsgaard EM, Husted SE. Improved nutritional status in elderly patients 6 months after stroke. J Nutr Health Aging. 2007 Jan-Feb;11(1):75-9. PMID 17315085
- [Result] Ekberg O, Hamdy S, Woisard V, Wuttge-Hannig A, Ortega P. Social and psychological burden of dysphagia: its impact on diagnosis and treatment. Dysphagia. 2002 Spring;17(2):139-46. doi: 10.1007/s00455-001-0113-5. PMID 11956839
- [Result] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Result] Wakabayashi H, Sakuma K. Rehabilitation nutrition for sarcopenia with disability: a combination of both rehabilitation and nutrition care management. J Cachexia Sarcopenia Muscle. 2014 Dec;5(4):269-77. doi: 10.1007/s13539-014-0162-x. Epub 2014 Sep 16. PMID 25223471
- [Result] Kuroda Y, Kuroda R. Relationship between thinness and swallowing function in Japanese older adults: implications for sarcopenic dysphagia. J Am Geriatr Soc. 2012 Sep;60(9):1785-6. doi: 10.1111/j.1532-5415.2012.04123.x. No abstract available. PMID 22985156
- [Result] Almirall J, Cabre M, Clave P. [Aspiration pneumonia]. Med Clin (Barc). 2007 Sep 29;129(11):424-32. doi: 10.1157/13110467. Spanish. PMID 17927938
- [Result] Germain I, Dufresne T, Gray-Donald K. A novel dysphagia diet improves the nutrient intake of institutionalized elders. J Am Diet Assoc. 2006 Oct;106(10):1614-23. doi: 10.1016/j.jada.2006.07.008. PMID 17000194
- [Result] Volkert D, Berner YN, Berry E, Cederholm T, Coti Bertrand P, Milne A, Palmblad J, Schneider S, Sobotka L, Stanga Z; DGEM (German Society for Nutritional Medicine); Lenzen-Grossimlinghaus R, Krys U, Pirlich M, Herbst B, Schutz T, Schroer W, Weinrebe W, Ockenga J, Lochs H; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Geriatrics. Clin Nutr. 2006 Apr;25(2):330-60. doi: 10.1016/j.clnu.2006.01.012. PMID 16735082
- [Result] Loeb MB, Becker M, Eady A, Walker-Dilks C. Interventions to prevent aspiration pneumonia in older adults: a systematic review. J Am Geriatr Soc. 2003 Jul;51(7):1018-22. doi: 10.1046/j.1365-2389.2003.51318.x. PMID 12834525
- [Result] Wieseke A, Bantz D, Siktberg L, Dillard N. Assessment and early diagnosis of dysphagia. Geriatr Nurs. 2008 Nov-Dec;29(6):376-83. doi: 10.1016/j.gerinurse.2007.12.001. PMID 19064135
- [Result] Cook IJ. Oropharyngeal dysphagia. Gastroenterol Clin North Am. 2009 Sep;38(3):411-31. doi: 10.1016/j.gtc.2009.06.003. PMID 19699405
- [Result] Hansen TS, Engberg AW, Larsen K. Functional oral intake and time to reach unrestricted dieting for patients with traumatic brain injury. Arch Phys Med Rehabil. 2008 Aug;89(8):1556-62. doi: 10.1016/j.apmr.2007.11.063. PMID 18674990
- [Result] Malone A, Hamilton C. The Academy of Nutrition and Dietetics/the American Society for Parenteral and Enteral Nutrition consensus malnutrition characteristics: application in practice. Nutr Clin Pract. 2013 Dec;28(6):639-50. doi: 10.1177/0884533613508435. Epub 2013 Oct 31. PMID 24177285
- [Result] Clave P, Shaker R. Dysphagia: current reality and scope of the problem. Nat Rev Gastroenterol Hepatol. 2015 May;12(5):259-70. doi: 10.1038/nrgastro.2015.49. Epub 2015 Apr 7. PMID 25850008

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who not agreed to participate or with severe oropharyngeal dysphagia (enteral feeding) was excluded
Period: Overall Study
Arm/Group | Modified Consistency and Volume Diet | Control Group
Started | 64 | 63
Completed | 54 | 51
Not Completed | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Consistency and Volume Diet | Control Group | Total
Number analyzed (Participants) | 54 | 51 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (10) | 71 (11) | 73 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 24 | 53
  Male | 25 | 27 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 51 | 105
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 54 | 51 | 105
Phase Angle (bioelectrical impedance) [Mean (Standard Deviation); unit: degrees] — This measurement was taken with a multifrequency bioelectrical impedance analyser (Inbody S10). The outcome is the result from the arctg X (resistance)/R (reactance)
  degrees | 4.4 (1.3) | 4.6 (1.4) | 4.5 (1.3)
Handgrip strength [Mean (Standard Deviation); unit: kg] | 15 (9) | 14 (10) | 15 (9)
Energy intake [Mean (Standard Deviation); unit: kcal/kg/d] | 27 (11) | 27 (10) | 27 (10)
Protein intake [Mean (Standard Deviation); unit: g/kg/d] | 1.3 (0.6) | 1.2 (0.5) | 1.3 (0.6)
Body weight [Mean (Standard Deviation); unit: kg] | 56 (12) | 56 (14) | 56 (14)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 21 (3.9) | 22 (5.0) | 21 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Adequacy of Oral Intake of Energy
Description: The energy intake measured in kcal/kg/d
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kcal/kg/d
Arm/Group | Modified Consistency and Volume Diet | Control Group
Number analyzed (Participants) | 54 | 51
kcal/kg/d | 41 (15) | 36 (12)

2. Primary Outcome: Adequacy of Oral Intake of Protein
Description: The protein intake measured in protein g/kg/d
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: g/kg/d
Arm/Group | Modified Consistency and Volume Diet | Control Group
Number analyzed (Participants) | 54 | 51
g/kg/d | 1.9 (0.68) | 1.5 (0.63)

3. Secondary Outcome: Body Weight
Description: The total of kg of body weight in the intervention group in contrast with the control group at 12 months of follow-up
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Modified Consistency and Volume Diet | Control Group
Number analyzed (Participants) | 54 | 51
kg | 62 (12) | 57 (15)

4. Secondary Outcome: Mortality
Description: number of deaths at 12 months of follow-up
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Consistency and Volume Diet | Control Group
Number analyzed (Participants) | 54 | 51
Participants | 8 | 18

5. Secondary Outcome: Swallowing Ability
Description: Patient's swallowing ability evaluated by volume-viscosity test, if patient is able to swallow correctly the three types of consistencies (liquid, nectar and pudding)
Time Frame: 12 months
Population: According to volume-viscosity test, number of patients that recovery the swallowing ability to eat safe
Measure: Number; unit: count of patients
Arm/Group | Modified Consistency and Volume Diet | Control Group
Number analyzed (Participants) | 54 | 51
count of patients | 26 | 22

6. Secondary Outcome: BMI
Description: Body mass index at the end of study
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Modified Consistency and Volume Diet | Control Group
Number analyzed (Participants) | 54 | 51
kg/m^2 | 24 (4.0) | 23 (6.0)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Modified Consistency and Volume Diet | Control Group
All-Cause Mortality (participants affected / at risk) | 8/54 | 18/51
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/51
Other Adverse Events (participants affected / at risk) | 0/54 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT02959450/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT02959450/SAP_001.pdf